CLINICAL TRIAL: NCT03441815
Title: A Double-blind, Randomized, Placebo-controlled Study of the Safety and Tolerability of Increasing Doses of XC8 After Single and Repeated Oral Administration in Healthy Volunteers
Brief Title: XC8 Safety, Tolerability and Pharmacokinetics in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: PHARMENTERPRISES LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: PULM-XC8-01
Record Dates: First submitted 2018-01-11; First posted 2018-02-22 (Actual); Last update posted 2018-02-22 (Actual); Status verified 2018-02

CONDITIONS: Asthma
Keywords: Healthy volunteers; Phase I; Histamine glutarimide; PHARMENTERPRISES
MeSH Terms: conditions — Asthma | interventions — histamine glutarimide

STUDY DESIGN:
Intervention Model Description: The dose cohorts were included into the study subsequently based on preliminary safety results evaluation performed by the Data Safety Monitoring Committee. 4 doses of XC8/placebo (2 mg, 10 mg, 50 mg and 200 mg) were used in the study.The duration of exposure to the study drug was 15 days in each cohort: Day 1, once, at the step of single administration, and then in 6 days, daily, 1 time a day for 14 days at the step of multiple administration.
Who Masked: Participant, Investigator
Masking Description: Blinding was carried out by using Placebo equivalent to XC8 tablets without active substance and the corresponding labeling of the study drug.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- XC8 2 mg (Experimental): Cohort 1: 6 subjects were randomized in a 2:1 ratio to be treated either with 2 mg XC8 (4 subjects) or placebo (2 subjects, see placebo arm).
  Interventions: Drug: XC8
- XC8 10 mg (Experimental): Cohort 2: 6 subjects were randomized in a 2:1 ratio to be treated either with 10 mg XC8 (4 subjects) or placebo (2 subjects, see placebo arm).
  Interventions: Drug: XC8
- XC8 50 mg (Experimental): Cohort 3: 6 subjects were randomized in a 2:1 ratio to be treated either with 50 mg XC8 (4 subjects) or placebo (2 subjects, see placebo arm).
  Interventions: Drug: XC8
- XC8 200 mg (Experimental): Cohort 4: 10 subjects were randomized in a 4:1 ratio to be treated either with 200 mg XC8 (8 subjects) or placebo (2 subjects, see placebo arm).
  Interventions: Drug: XC8
- Placebo (Placebo Comparator): Placebo comparator arm consists of 8 subjects (2 subjects in each cohort).
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: XC8
  Other Names: Histamine glutarimide
  Arms: XC8 10 mg; XC8 2 mg; XC8 200 mg; XC8 50 mg
Drug: Placebo
  Arms: Placebo

SUMMARY:
A double-blind, randomized, placebo-controlled, Phase I clinical study of the safety and tolerability of increasing doses of XC8 after single and repeated oral administration in healthy volunteers. The volunteers received the study drug once, and then continued daily intake for 14 days after a 6-day break.

The primary objective of the study was to evaluate the safety and tolerability profile for XC8 after single and multiple administration based on the frequency and severity of adverse events and changes in vital signs, laboratory results, electrocardiography and results of the physical examination.

The secondary objective of the study was to assess pharmacokinetics of XC8.

DETAILED DESCRIPTION:
One Russian center was approved for participation in this study. One center was initiated. Healthy volunteers were enrolled in 1 center. The study consisted of 4 periods: screening, single administration, multiple administration and follow-up.

All eligible subjects were randomized into the study in appropriate cohort groups sequentially.

Cohort 1 - XC8 or Placebo 2 mg once and then daily 14 days after a 6-day break; Cohort 2 - XC8 or Placebo 10 mg once and then daily during 14 days after a 6-day break; Cohort 3 - XC8 or Placebo 50 mg once and then daily during 14 days after a 6-day break; Cohort 4 - XC8 or Placebo 200 mg once and then daily during 14 days after a 6-day break.

The decision regarding increasing of the study drug dose for a subsequent cohort was made by the Data Safety Monitoring Committee on the basis of preliminary safety results assessment.

A total of 20 volunteers received XC8 (2 mg, 10 mg, 50 mg or 200 mg) and a total of 8 volunteers received the placebo during the study participation. The follow-up period lasted for 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Non-smoking men aged 18 to 50 years (inclusive);
2. Verified diagnosis "healthy" according to standard clinical, laboratory and instrumental methods of examination;
3. Body mass index of 19 to 30 kg/m2 (inclusive);
4. Consent to use reliable methods of contraception during the study and 3 months after its completion (condoms with spermicide);
5. Signed patient information sheet and informed consent form for participation in the study.

Exclusion Criteria:

1. Hepatic disorder or renal disease; any other disease that, in the opinion investigator, may affect the results of the study, or may lead to the health aggravation during the study;
2. Laboratory abnormalities at screening;
3. Course intake of medicinal products (including herbs and biologically active additives) for preventive or curative purposes within 1 month prior to screening;
4. Antibodies to HIV and hepatitis C virus, the presence of the hepatitis B surface antigen, a positive syphilis test;
5. The presence of a sleep disorder (for example, night work, sleep disturbances, insomnia, recent return from another time zone, etc.);
6. Signs of alcohol or drug abuse; taking alcohol or drugs during 4 days before screening;
7. History of allergies (including medicines and food products);
8. Symptomatic rhinitis in anamnesis during 2 years prior to screening (allergic rhinitis, non-allergic rhinitis or pollinosis);
9. Blood donation / plasma, surgical intervention (in a hospital environment) during 12 weeks before screening;
10. Participation in other clinical trials or taking the study drug during 3 months before screening;
11. Impossibility to understand or follow protocol instructions;
12. Smoking 3 months before screening;
13. Lactase deficiency, lactose intolerance, glucose-galactose malabsorption;
14. Acute infectious diseases less than 4 weeks before the start of the study.

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2015-02-14 (Actual); Primary Completion 2015-07-07 (Actual); Study Completion 2015-07-07 (Actual)

PRIMARY OUTCOMES:
Number of Adverse events per treatment arm | Change from pre-dose to Day 50
  Adverse events will be summarized descriptively by treatment arm. Verbatim terms will be mapped to preferred terms and organ systems using the current Medical Dictionary for Regulatory Activities version. For each preferred term, frequency counts and percentages will be calculated by cohort.The nature, severity, seriousness, and relationship to study medication will be summarized for all study subjects
Physical examination | Day 1 till Day 36
  Physical examination results will be listed for following: general appearance, skin, head, eyes, ears, nose, throat, neck (including thyroid), lymph nodes, chest, heart, abdomen (including liver examination), extremities, and nervous system.
12-lead ECG | Change from pre-dose till Day 36
  12-lead ECG results will be analyzed descriptively

SECONDARY OUTCOMES:
Pharmacokinetics of XC8 by assessing AUC0-inf | Day 1 and 21 (Pre dose, and 20 min, 40 min, 1, 2, 4, 6 and 10 hours post dose), Day 2 and Day 22 (24 hours ±10 minutes post dose), Day 3 (48 hours ±10 minutes post dose), Day 4 (72 hours ±10 minutes post dose), Day 8 to 12 and 15 (Pre dose)
  Area under the curve "concentration of the drug-time" from the time of administration of the drug till infinity
Pharmacokinetics of XC8 by assessing Cmax | Day 1 and 21 (Pre dose, and 20 min, 40 min, 1, 2, 4, 6 and 10 hours post dose), Day 2 and Day 22 (24 hours ±10 minutes post dose), Day 3 (48 hours ±10 minutes post dose), Day 4 (72 hours ±10 minutes post dose), Day 8 to 12 and 15 (Pre dose)
  Maximum plasma concentration
Pharmacokinetics of XC8 by assessing AUC0-t | Day 1 and 21 (Pre dose, and 20 min, 40 min, 1, 2, 4, 6 and 10 hours post dose), Day 2 and Day 22 (24 hours ±10 minutes post dose), Day 3 (48 hours ±10 minutes post dose), Day 4 (72 hours ±10 minutes post dose), Day 8 to 12 and 15 (Pre dose)
  Area under the curve "concentration of the drug-time" from the time of administration of the drug till the time (t) the last blood sampling
Pharmacokinetics of XC8 by assessing Tmax | Day 1 and 21 (Pre dose, and 20 min, 40 min, 1, 2, 4, 6 and 10 hours post dose), Day 2 and Day 22 (24 hours ±10 minutes post dose), Day 3 (48 hours ±10 minutes post dose), Day 4 (72 hours ±10 minutes post dose), Day 8 to 12 and 15 (Pre dose)
  Time to maximum drug concentration in the blood plasma administration
Pharmacokinetics of XC8 by assessing T1/2 | Day 1 and 21 (Pre dose, and 20 min, 40 min, 1, 2, 4, 6 and 10 hours post dose), Day 2 and Day 22 (24 hours ±10 minutes post dose), Day 3 (48 hours ±10 minutes post dose), Day 4 (72 hours ±10 minutes post dose), Day 8 to 12 and 15 (Pre dose)
  Terminal elimination half-life
Pharmacokinetics of XC8 by assessing kel | Day 1 and 21 (Pre dose, and 20 min, 40 min, 1, 2, 4, 6 and 10 hours post dose), Day 2 and Day 22 (24 hours ±10 minutes post dose), Day 3 (48 hours ±10 minutes post dose), Day 4 (72 hours ±10 minutes post dose), Day 8 to 12 and 15 (Pre dose)
  Elimination rate constant
Pharmacokinetics of XC8 by assessing Cav | Day 8 to 12 and 15 (Pre dose); Day 21 (Pre dose, and 20 min, 40 min, 1, 2, 4, 6 and 10 hours post dose), Day 22 (24 hours ±10 minutes post dose
  Average concentration over one dosing interval

CONTACTS AND LOCATIONS:
Locations (1):
- SBEI HPE The First Moscow State Medical University n.a. Sechenov of Ministry of Health of Russian Federation, University Hospital #2, Department of Development of New Medicines, Moscow, Russia

IPD SHARING:
Plan to Share IPD: No